CLINICAL TRIAL: NCT06217068
Title: Comparative Analysis of Biomarkers in Physically Active and Sedentary College Students
Brief Title: Comparative Analysis of Biomarkers in Response to Acute Moderate-Intensity Activity
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Jennifer Gay, Associate Professor, University of Georgia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PROJECT00008178
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Acute Exercise; Aerobic Exercise; Biomarkers

STUDY DESIGN:
Intervention Model Description: Two group pre-test post-test study where groups are determined by current activity level (sedentary versus active). The dose of exercise is being tested between groups to see if there are differential effects of this acute dose at this intensity on biomarkers.
Who Masked: Outcomes Assessor
Masking Description: Lab processing the blood samples is blinded to participant group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sedentary Individuals - Acute Moderate-Intensity Exercise (Experimental): 8 minutes of elliptical exercise at a moderate intensity based on heart rate reserve. There will be a 2-minute warm-up and 2-minute cool down period in addition to the 8 minutes at moderate-intensity.
  Interventions: Behavioral: Elliptical Activity
- Active Individuals - Acute Moderate-Intensity Exercise (Experimental): 8 minutes of elliptical exercise at a moderate intensity based on heart rate reserve. There will be a 2-minute warm-up and 2-minute cool down period in addition to the 8 minutes at moderate-intensity.
  Interventions: Behavioral: Elliptical Activity

INTERVENTIONS:
Behavioral: Elliptical Activity — 8 minutes of elliptical exercise at a moderate intensity based on heart rate reserve. There will be a 2-minute warm-up and 2-minute cool down period in addition to the 8 minutes at moderate-intensity.

SUMMARY:
The purpose of this study is to understand how college students' biomarkers change with a relatively short bout of moderate-intensity physical activity. The investigators are comparing biomarkers in between self-reported physically active and sedentary students in terms of their percent difference and change. The investigators are also studying physically active versus sedentary college students' mental health. This is a mentored student research project in the investigator's lab (not part of a thesis, dissertation, or other coursework requirements), where multiple students have developed research questions using the same study design.

DETAILED DESCRIPTION:
This study will use a two-group (sedentary versus active) pre-test, post-test study design. Following the informed consent process, participants will complete the pre-test data collection protocol including the first venipuncture blood draw for ammonia, insulin, cortisol, and c-reactive protein, first finger stick blood sample for glucose measurement, reporting of food eaten for the day as well as transportation methods to the study site. Resting heart rate will be measured.

Following a 15-minute waiting period to minimize potential effects from the blood draw, participants will walk with a study team member to a reserved elliptical machine. For the exercise component, the lab member will emphasize to the participant about maintaining the desired heart rate for moderate intensity exercise. The participant will use the elliptical for 12 minutes, without music, conversation, or general entertainment. Appropriate warm-up and cool-down is added in to the exercise time (the first two minutes and last two minutes) with preference of moderate intensity exercise lasting 8 minutes.

Participants will then walk with the study team member back to the Lab for post-test data collection. Post-test data collection follows the same procedures as pre-test data collection. Participants also will take a mental health questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* This study will enroll full-time students at the investigator's university who are aged 18-34 years.
* Participants will be generally healthy participants, assessed using the 2020 Physical Activity Readiness Questionnaire (first 7 questions) as a screening tool. Individuals who answer "no" to all of the 7 questions will be deemed healthy enough to take part.
* Two balanced groups will be created based on self-reported current activity level, either sedentary (<30min/week of exercise) or meeting exercise guidelines (>=150min/week of exercise).
* Potential participants should be willing to complete the blood draws and the 12 minutes of moderate-intensity exercise on an elliptical machine.
* Potential participants should be able to speak and read the English language. This is so they will be able to understand the study protocols clearly.

Exclusion Criteria:

* Are allergic to nuts because the snacks provided following the blood draw may contain nut products.
* Do not have transportation and parking (if needed) to lab.

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Ammonia | Pre-test and post-test (immediately following exercise)
  Blood sample
Insulin | Pre-test and post-test (immediately following exercise)
  Blood sample
Cortisol | Pre-test and post-test (immediately following exercise)
  Blood sample
C-reactive protein | Pre-test and post-test (immediately following exercise)
  Blood sample
Glucose | Pre-test and post-test (immediately following exercise)
  Blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Gay, PhD, Principal Investigator — University of Georgia
Locations (1):
- University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
We do not anticipate sharing individual, identified data to other researchers.